CLINICAL TRIAL: NCT00445406
Title: Bevacizumab and Pegylated Liposomal Doxorubicin as First-Line Therapy for Locally Recurrent or Metastatic Breast Cancer. A Multicenter, Single-Arm Phase II Trial
Brief Title: Bevacizumab and Doxorubicin Hydrochloride Liposome in Treating Women With Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 24/06; EU-20701
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bevacizumab + doxorubin hydrochloride liposme — Patients receive bevacizumab IV over 30-90 minutes and doxorubicin hydrochloride liposome IV over 30-90 minutes on days 1 and 15. Treatment repeats every 4 weeks for up to 6 courses
Drug: Bevacizumab — Patients then receive bevacizumab alone IV over 30-90 minutes on days 1 and 15. Courses with bevacizumab repeat every 4 weeks in the absence of disease progression or unacceptable toxicity

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab also may stop the growth of breast cancer by blocking blood flow to the tumor. Drugs used in chemotherapy, such as doxorubicin hydrochloride liposome, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with doxorubicin hydrochloride liposome may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving bevacizumab together with doxorubicin hydrochloride liposome works in treating women with locally recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability of bevacizumab and doxorubicin hydrochloride liposome in women with locally recurrent or metastatic breast cancer.

Secondary

* Determine the efficacy of this regimen in these patients.
* Identify surrogate markers of angiogenesis, including vascular endothelial growth factor (VEGF), VEGF receptor 1, and matrix metalloproteinase 9, in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive bevacizumab IV over 30-90 minutes and doxorubicin hydrochloride liposome IV over 30-90 minutes on days 1 and 15. Treatment repeats every 4 weeks for up to 6 courses*. Patients then receive bevacizumab alone IV over 30-90 minutes on days 1 and 15. Courses with bevacizumab repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients may receive additional courses of doxorubicin hydrochloride liposome at the discretion of the primary investigator.

Blood samples are collected at baseline, on day 1 of course 3 and then once every 3 months during study treatment, and after completion of study treatment. Samples are analyzed by enzyme-linked immunosorbent assay to determine the level of circulating angiogenesis-related molecules, including serum vascular endothelial growth factor (VEGF), VEGF receptor 1, and matrix metalloproteinase 9.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 43 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically or histologically confirmed breast cancer

  * Metastatic OR locally recurrent disease
  * Unresectable disease
  * Not amenable to radiotherapy
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan

  * Measurable disease must be outside irradiated areas
* ErbB2-negative disease by immunohistochemistry (negative or 1+) or fluorescent in situ hybridization (FISH)
* No known CNS metastases, even if previously treated
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* WHO performance status 0-1
* LVEF ≥ 55%
* Hemoglobin ≥ 10.0 g/dL
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin < 2 times upper limit of normal (ULN)
* ALT ≤ 2.5 times ULN (5 times ULN if liver metastases are present)
* Alkaline phosphatase (AP) ≤ 2.5 times ULN

  * AP > 2.5 times ULN and ≤ 6 times ULN allowed if ALT ≤ 1.5 times ULN
  * AP > 6 times ULN allowed if ALT normal
* Creatinine ≤ 1.5 times ULN
* Proteinuria < 2+ by dipstick OR protein ≤ 1 g/24hr-urine collection
* INR ≤ 1.5 OR Quick ≥ 70%
* aPTT ≤ 1.5 times ULN
* No peripheral neuropathy > grade 2
* No history or evidence of hereditary bleeding diathesis or coagulopathy with the risk of bleeding
* No uncontrolled hypertension, defined as systolic blood pressure (BP) > 150 mm Hg and/or diastolic BP > 100 mm Hg, measured repeatedly at > 2 visits despite adequate treatment with ≥ 2 different antihypertensive drugs
* No clinically significant cardiovascular disease, including the following:

  * Cerebrovascular accident or stroke within the past 6 months
  * Myocardial infarction within the past 6 months
  * Unstable angina
  * New York Heart Association class II-IV congestive heart failure
  * Serious cardiac arrhythmia (e.g., ventricular arrhythmia, high-grade atrioventricular-block) not controlled by medication or requiring medication which might interfere with regularity of the study treatment
* No serious nonhealing wound, active peptic ulcer, nonhealing bone fracture, or bleeding skin metastases
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No active infection requiring IV antibiotics
* No known hypersensitivity to any of the study drugs or excipients
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* No evidence of any other disease that contraindicates the use of an investigational drug, that may affect patient compliance with study routines, or places the patient at high risk for treatment-related complications including, but not limited to, the following:

  * Metabolic dysfunction
  * Physical examination finding
  * Psychological dysfunction
  * Clinical laboratory finding giving reasonable suspicion of a disease or condition
* No known CNS disease unrelated to cancer (e.g., uncontrolled seizures), unless adequately treated with standard medical therapy
* No high-risk factors for bleeding, including the following:

  * Coagulation parameters outside range
  * Need for concurrent anticoagulant therapy
  * Insufficient time gap after surgical procedures
* No other malignancy within the past 5 years except for adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* No significant traumatic injury within the past 28 days
* No known HIV positivity
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study therapy

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for metastatic or inoperable locally recurrent breast cancer
* No prior bevacizumab or other anti-vascular endothelial growth factor drug therapy
* No prior radiotherapy involving the heart (usual irradiation dose to breast or chest wall allowed)
* More than 12 months since prior neoadjuvant or adjuvant chemotherapy
* No neoadjuvant or adjuvant doxorubicin hydrochloride with cumulative dose > 360 mg/m² or epirubicin hydrochloride with cumulative dose > 720 mg/m²
* More than 6 months since prior adjuvant radiotherapy
* More than 28 days since prior major surgical procedure with high risk of bleeding
* More than 24 hours since prior minor surgical procedures
* More than 10 days since prior acetylsalicylic acid (> 325 mg/day) or clopidogrel bisulfate (> 75 mg/day)
* More than 10 days since prior and no concurrent use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes

  * Prophylactic use of anticoagulants allowed (e.g., for maintenance of venous catheter)
* More than 30 days since prior investigational therapies or participation in other investigational studies
* No concurrent hormonal therapy
* No other concurrent antineoplastic or antitumor therapy
* No other concurrent investigational drugs
* No concurrent radiotherapy
* No concurrent nonsteroidal anti-inflammatory drugs with activity on platelets and gastric mucosa (e.g., dipyridamole, clopidogrel bisulfate, acetylsalicylic acid)
* No anticipated need for major surgery during the course of the study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-12; Primary Completion 2008-09 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
bevacizumab and doxorubicin hydrochloride liposome | Until treatment ends
  Determine the safety and tolerability of bevacizumab and doxorubicin hydrochloride liposome.

SECONDARY OUTCOMES:
Determine the efficacy of this regimen | Until treament ends
  Determine the efficacy of this regimen in these patients.
Identify surrogate markers of angiogenesis | Until treatment ends
  Identify surrogate markers of angiogenesis, including vascular endothelial growth factor (VEGF), VEGF receptor 1, and matrix metalloproteinase 9, in patients treated with this regimen.
Overall (complete and partial) response as measured by RECIST criteria | Periodically
Time to treatment failure | Until treatment ends
Progression-free survival | Periodically
Overall survival | Life-long

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Rochlitz, MD, Study Chair — Universitaetsspital-Basel
Locations (1):
- Universitaetsspital-Basel, Basel, Switzerland

REFERENCES:
- [Result] Rochlitz C, Ruhstaller T, Lerch S, Spirig C, Huober J, Suter T, Buhlmann M, Fehr M, Schonenberger A, von Moos R, Winterhalder R, Rauch D, Muller A, Mannhart-Harms M, Herrmann R, Cliffe B, Mayer M, Zaman K; Swiss Group for Clinical Cancer Research (SAKK). Combination of bevacizumab and 2-weekly pegylated liposomal doxorubicin as first-line therapy for locally recurrent or metastatic breast cancer. A multicenter, single-arm phase II trial (SAKK 24/06). Ann Oncol. 2011 Jan;22(1):80-85. doi: 10.1093/annonc/mdq319. Epub 2010 Jul 1. PMID 20595448